CLINICAL TRIAL: NCT02882412
Title: Effectiveness of Buprenorphine/Naloxone in Patients With Chronic Pain and Iatrogenic Opioid Dependence
Brief Title: Effectiveness of Buprenorphine/Naloxone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1551
Record Dates: First submitted 2016-08-04; First posted 2016-08-29 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Chronic Pain
Keywords: effectiveness; buprenorphine/naloxone; iatrogenic opioid dependence
MeSH Terms: conditions — Chronic Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient group
  Interventions: Other: observational

INTERVENTIONS:
Other: observational

SUMMARY:
Long-term use of opioids for chronic pain is a growing health and social problem, mainly because of the risk of dependence. Buprenorphine/naloxone is used as substitution therapy for opioid dependence. This substitution therapy in patients with opioid dependence lessens withdrawal symptoms and craving. There is limited research on the effectiveness of buprenorphine/naloxone in patients with chronic pain and iatrogenic opioid dependence. The primary aim of this study is to investigate the effectiveness of buprenorphine/naloxone in patients suffering from chronic pain and an iatrogenic induced dependence on opioids. This study will investigate the effects of opioid substitution by buprenorphine/naloxone in patients suffering from chronic pain using long-term opioids, with pain and withdrawal symptoms as primary outcome measures. Secondary outcome measures will be craving, substance use, psychiatric comorbidity and quality of life.

DETAILED DESCRIPTION:
This is a prospective open-label observational cohort study (exploratory pilot). Investigators will include 20 patients between 18 and 65 years with chronic pain and dependence on opioids, who were referred by their physician for replacement of opioids to buprenorphine/naloxone. Exclusion criteria are contraindications for buprenorphine/naloxone and patients with psychiatric disorders requiring acute treatment. The degree of pain and withdrawal symptoms will be assessed by the Quantitative Sensory Testing (QST) measurement and the following questionnaires: Visual Analog Scale (VAS), Objective Withdrawal Scale (OWS) and Subjective Withdrawal Scale (SWS). Secondary, craving and substance use/degree of opioid dependence will be studied using the Current Opioid Misuse Measure (COMM) and Obsessive Compulsive Drug using Scale (OCDS). Psychiatric comorbidity will be assessed using the following questionnaires: Depression, Anxiety and Stress Scale (DASS), Personality Inventory for DSM-5 (PID 5-BF), The 20-item Toronto Alexithymia Scale (TAS-20), Inventory of Depressive Symptomatology (IDS), the Perseverative Thinking Questionnaire (PTQ) and Mini International Neuropsychiatric Interview (MINI). These questionnaires are part of the standard assessment at the department of psychiatry at the Radboud University Medical Centre, Nijmegen. The EuroQol five dimensions questionnaire (EQ5D) will be used to assess the quality of life. During the replacement of opioids to buprenorphine/naloxone, the buprenorphine/naloxone protocol will be used.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged 18 to 65 years
* suffering from chronic pain (pain for more than 6 months)
* iatrogenic opioid dependence (according to the DSM-5 criteria)
* there is informed consent for using the data for scientific analyses.

Exclusion Criteria:

* Contraindications for buprenorphine/naloxone, such as severe respiratory insufficiency, severe hepatic insufficiency, alcohol intoxication or delirium tremens.
* In addition participants with psychiatric disorders requiring acute treatment will be excluded, for instance an acute psychosis, acute manic episode or patients who are suicidal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women aged 18 to 65 years suffering from chronic pain (pain for more than 6 months) and iatrogenic opioid dependence (according to the DSM-5 criteria).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Pain with QST baseline and change from baseline from QST at 2 months | baseline and change from baseline from QST at 2 months
  QST: Quantitative Sensory Testing
withdrawal symptoms | baseline and change from baseline from OWS at 2 months
  OWS: Objective Withdrawal Scale
Pain with VAS baseline and change from baseline from QST at 2 months | baseline and change from baseline from VAS at 2 months
  VAS: Visual Analogue Scale
withdrawal symptoms | baseline and change from baseline from SWS at 2 months
  SWS: Subjective Withdrawal Scale

SECONDARY OUTCOMES:
psychiatric comorbidity | baseline and change from baseline from DASS at 2 months
  DASS: Depression Anxiety Stress Scale
psychiatric comorbidity | baseline and change from baseline from MINI at 2 months
  MINI: Mini International neuropsychiatric Interview
craving | baseline and change from baseline from OCDS at 2 months
  OCDS: Obsessive Compulsive Drug using Scale
degree of opioids dependence | baseline and change from baseline from COMM at 2 months
  COMM: Current Opioid Misuse Measure
psychiatric comorbidity | baseline and change from baseline from PID-5-BF at 2 months
  PID-5-BF: Personality Inventory for DSM-5
psychiatric comorbidity | baseline and change from baseline from TAS-20 at 2 months
  TAS-20: the 20-item Toronto Alexithymia Scale
psychiatric comorbidity | baseline and change from baseline from IDS at 2 months
  IDS: Inventory of Depressive Symptomatology
psychiatric comorbidity | baseline and change from baseline from PTQ at 2 months
  PTQ: The Perseverative Thinking Questionnaire
Quality of life with EQ5D baseline and change from baseline from EQ5D at 2 months | baseline and change from baseline from EQ5D at 2 months
  EQ5D: EuroQol five dimensions questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Arnt Schellekens, Phd, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided